CLINICAL TRIAL: NCT05699083
Title: Evaluation of Patient Reported Outcomes After Weight Loss Surgery in Low-Risk Patients
Brief Title: Outcomes After Weight Loss Surgery in Low-Risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Feiz & Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MF001
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Weight Loss; Bariatric Surgery
Keywords: Outcomes
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Pre-post interventional study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with BMI between 30-34.5 kg/m2 (Other): Patients with BMI between 30-34.5 kg/m2 will be administered a body image/self-esteem questionnaire pre-operatively and at 1 month, 3 months, 6 months and 12 months post-operatively.
  Interventions: Other: Body Image/Self-Esteem Questionnaires

INTERVENTIONS:
Other: Body Image/Self-Esteem Questionnaires — Pre-operation and post-operation questionnaires to assess factors including but not limited to body image, quality of life, and self-esteem.

SUMMARY:
The purpose of this research is to determine patient-reported outcomes after weight loss surgery, including changes in health, mood, quality of life, health satisfaction, and emotional health, in low-risk patients. Weight loss surgery has been well studied for patients with body mass index (BMI) 35 kg/m^2 or more and those with weight-related medical problems who have a BMI 30 kg/m^2 or more. However, outcomes after weight loss surgery in patients with BMI under 35 kg/m^2 and without co-morbidities have not been well studied.

DETAILED DESCRIPTION:
The purpose of this research is to determine patient-reported outcomes after weight loss surgery in low-risk patients. Weight loss surgery has been well-studied for patients with body mass index (BMI) 35 kg/m^2 or more and those with weight-related medical problems who have a BMI 30 kg/m^2 or more. Weight-related medical problems, also called co-morbidities, can include diabetes mellitus, hypertension, sleep apnea, and degenerative joint diseases. The surgery is considered safe and effective. Outcomes after weight loss surgery in patients with BMI under 35 kg/m^2 and without co-morbidities have not been well studied. The investigators' purpose is to study patient-reported outcomes after weight loss surgery in patients with BMI between 30 kg/m^2 and 34.5 kg/m^2 without co-morbidities. These include changes in health, mood, quality of life, health satisfaction, and emotional health.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI between 30 kg/m2 and 34.5 kg/m2 without co-morbidities who are medically cleared to undergo cosmetic weight loss surgery.
* Written informed consent obtained from the subject or the subject's legal representative and the ability for the subject to comply with the requirements of the study.

Exclusion Criteria:

* Patients who are pregnant.
* Patients with BMI below 30 kg/m2.
* Patients with BMI above 34.5 kg/m2.
* Patients who have co-morbidities including, but not limited to, diabetes mellitus, hypertension, sleep apnea, and degenerative joint disease.
* Patients who are not medically cleared to undergo weight loss surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-01-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Change in Perception of General Health | 0, 1, 3, 6, 12 months
  A survey will be administered to determine changes in one's self-assessed general health.
Change in Perception of Body Image | 0, 1, 3, 6, 12 months
  Surveys will be administered to determine changes in one's self-assessed body image.
Change in Perception of Quality of Life | 0, 1, 3, 6, 12 months
  Surveys will be administered to determine changes in one's self-assessed quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Feizbakhsh, MD, Principal Investigator — Dr. Feiz and Associates
Locations (1):
- Dr. Feiz and Associates, Beverly Hills, California, United States